CLINICAL TRIAL: NCT05922176
Title: Biomarker Screening for Immunotherapy Response Evaluation Using Microneedle Patch in Patients with Allergic Rhinitis
Acronym: MIST
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Park Kyung Hee, Clinical Associate Professor, Yonsei University
Other Study IDs: 4-2023-0353
Record Dates: First submitted 2023-06-18; First posted 2023-06-28 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, skin tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patient group of House dust mist allergic rhinitis: 1. Adult male and female patients aged 19 to 60 with allergic rhinitis caused by the antigen of the American house dust mite (It is judged that the positive for the house dust mite is MAST ≥ Class 3 or ImmunoCAP® ≥3.5 kUA/L)
  2. Moderate-severe persistent rhinitis when evaluated according to ARIA (Allergic rhinitis and its impact on asthma)
  3. A person who has signed a written consent to participate in this clinical trial at his/her own discretion after fully explaining the purpose, contents, characteristics of the test drug, and expected adverse reactions prior to participation in the clinical trial
  Interventions: Other: Evaluation of clinical indicators, Sample collection before& after immunotherapy
- control group: 1. Adults 19 years of age or older who are judged to be free from skin diseases or allergic diseases through medical examination and visual observation by a specialist
  2. A person who agrees to provide samples derived from the human body
  3. A person who voluntarily agreed to this study and prepared a consent form after approval of the IRB
  Interventions: Other: Sample collection before& after immunotherapy

INTERVENTIONS:
Other: Evaluation of clinical indicators, Sample collection before& after immunotherapy — A. Evaluation of clinical indicators before immunotherapy
  1. Symptom Scale for Rhinitis: Total Nasal Symptom Score (TNSS), Rhnitis Quality of Life Questionnaire(RQLQ)
  2. American house dust mite-specific immunogloblin G4 (sIgG4)
  3. American house dust mite-specific immunogloblin E (sIgE)
  B. Sample collection before immunotherapy
  1. Skin: Skin test using minimally invasive microstructure patch stripping method
  2. Blood: Measurement of blood immunological indicators (Th2, Treg-related cytokine and blocking factor, etc.)
  C. Evaluation of clinical indicators 4 to 6 months after immunotherapy
  : Treatment is performed for about 4 months, and the progress of treatment is evaluated through the evaluation of the following clinical indicators.
  same as examination in 'A'
  D. Sample collection after 4 to 6 months of immunotherapy same as examination in 'B'
  Groups: patient group of House dust mist allergic rhinitis
Other: Sample collection before& after immunotherapy — B. Sample collection before immunotherapy
  1. Skin: Skin test using minimally invasive microstructure patch stripping method
  2. Blood: Measurement of blood immunological indicators (Th2, Treg-related cytokine and blocking factor, etc.)
  D. Sample collection after 4 to 6 months of immunotherapy
  1. Skin: Skin test using minimally invasive microstructure patch stripping method
  2. Blood: Measurement of blood immunological indicators (Th2, Treg-related cytokine and blocking factor, etc.)
  Groups: control group

SUMMARY:
Allergic rhinitis is a disease in which the nasal mucous membrane overreacts to allergens, resulting in symptoms such as spasmodic and repetitive sneezing, rhinorrhea, and stuffy nose, and can be treated with immunotherapy for radical treatment. Immunotherapy treatments include subcutaneous injections, sublingual tablets, and sublingual fluids, and subcutaneous injections have the risk of anaphylaxis, the hassle of daily administration at home, and local allergic reactions. Transdermal absorption immunotherapy (DF19001) that can compensate for the shortcomings of these existing immunotherapy drugs is currently under clinical research in Korea (Severance Hospital IRB No. 4-2021-1345).

Immunotherapy requires periodic monitoring, such as analyzing immunological changes through sample collection and determining the dose and cycle of administration, because the treatment period is long and individual immune responses are different. Existing methods for confirming immune responses in samples used invasive skin biopsy and blood collection methods, but in-blood evaluation indicators have the disadvantage of being ineffective as initial efficacy evaluations or predictive evaluations before treatment. In addition, skin biopsy should be performed by a specialist, and there is a disadvantage that resistance occurs because the patient's pain is accompanied, and scars or bruises may remain. Therefore, since it is a biopsy through minimal invasion compared to a tissue biopsy, the investigators would like to use a method of collecting skin samples through a microstructure (micro needle patch), a method that has little pain and no scars. Through this study, RNA is obtained from patients with house dust mite allergic rhinitis through minimally invasive skin samples, and immunotherapy response evaluation biomarkers are screened according to immunotherapy implementation, and its use as an indicator of immunotherapy prognosis in allergic diseases.

DETAILED DESCRIPTION:
Allergic rhinitis is a disease in which the nasal mucosa overreacts to allergens, resulting in symptoms such as seizure and repetitive sneezing, runny nose, and stuffy nose. Typical treatments include avoiding causative substances and anti-allergic medication. Immunotherapy may not be sufficient for treatment satisfaction with existing treatments, it is practically impossible to avoid allergens, or allergen specific immunotherapy may be performed for more root treatment.

Immunotherapy is known as the only way to change the natural course of allergic diseases by increasing the amount of substances that cause allergic reactions to allergic patients from a small amount and reducing allergic reactions through repeated administration for three to five years. Immunotherapy treatments include hypodermic injections, hypodermic tablets, and hypodermic fluids, and each has its pros and cons. Subcutaneous injection immunotherapy requires regular visits to a medical institution for injection, and there is a risk of anaphylaxis. Although sublingual immunotherapy has a low risk of anaphylaxis, it is cumbersome to administer it daily at home, and the incidence of local allergic reactions in the oral cavity is high due to 30 to 70 times less absorption in the body than injection treatments. Transdermal absorption immunotherapy (DF19001) that can compensate for the shortcomings of these existing immunotherapy drugs is currently under clinical research in Korea (Serbans Hospital IRB No. 4-2021-1345).

These immunotherapy require periodic monitoring, such as analyzing immunological changes through sample collection and determining administration dose and cycle, because the treatment period is long at 3-5 years and individual immune responses are different. Most of the existing methods for confirming immune responses in samples used invasive skin biopsy or blood collection methods, but allergen specific IgE (allergen specific IgG4, blocking factors) have the disadvantage of being ineffective as an initial efficacy evaluation or a pre-treatment prediction evaluation of a subject. In addition, various analysis methods can be used through skin biopsy to see changes in the initial immune response of the inoculation site, but this must be performed by a specialist, and has the disadvantage of being resistant to patient pain and scarring or bruising.

Therefore, in order to overcome these difficulties through this clinical study, the investigators would like to use a method of collecting skin samples through a microstructure (micro needle patch). When the microstructure patch is applied to the skin surface for 5 minutes, it passes through the microstructure's fine needle (<0.5 mm long) keratin layer and enters the inside of the skin as shown in the image below. Various immunological indicators are analyzed by collecting skin factors remaining in the patch by applying the patch for a sufficient time for various factors in the epidermis and dermis layer to be adsorbed through the microstructure that has entered the skin.

Since this method is a biopsy through minimal invasion compared to conventional tissue biopsy, there is little pain and no scarring, and previous studies have confirmed that a small amount of RNA can be separated from skin samples using microstructure patches and microarray can be performed. In addition, in the same way, the detection of protein biomarkers according to the test collection method for determining treatment in patients with atopic dermatitis was observed.

Therefore, this study aims to obtain RNA from patients with house dust mite allergic rhinitis through minimally invasive skin samples, screen the biomarker for immunotherapy response evaluation through immunotherapy and confirm its use as an indicator of immunotherapy prognosis in allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* A. patient group of House dust mite

  1. Adult male and female patients aged 19 to 60 with allergic rhinitis caused by the antigen of the American house dust mite (It is judged that the positive for the house dust mite is MAST ≥ Class 3 or ImmunoCAP® ≥3.5 kUA/L)
  2. Moderate-severe persistent rhinitis when evaluated according to ARIA (Allergic rhinitis and its impact on asthma)
  3. A person who has signed a written consent to participate in this clinical trial at his/her own discretion after fully explaining the purpose, contents, characteristics of the test drug, and expected adverse reactions prior to participation in the clinical trial B. Control group (Normal person)

  <!-- -->

  1. Adults 19 years of age or older who are judged to be free from skin diseases or allergic diseases through medical examination and visual observation by a specialist
  2. A person who agrees to provide samples derived from the human body
  3. A person who voluntarily agreed to this study and prepared a consent form after approval of the IRB

Exclusion Criteria:

* A. patient group of House dust mite

  1. Patients who are taking drugs that may affect efficacy evaluation (but can participate if there is no change in the drug taken during the study period)
  2. Within six months of participation in the study, other clinical trial drugs or biological equivalence test drugs, biological agents (e.g. Anti-IgE) were administered
  3. If there is a skin disease or tattoo in the area where the medication is applied
  4. Immunosuppressive therapy or systemic steroid therapy for acute and chronic inflammatory skin diseases
  5. A person in charge of testing or a person in charge of testing deemed inappropriate to participate in the test due to other reasons B. Control (Normal person)

  <!-- -->

  1. Patients with allergic diseases such as atopic dermatitis or allergic asthma and rhinitis
  2. A person who voluntarily disagrees with this study after approval of the IRB and has not completed the consent form

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Adult male and female patients aged 19 to 60 with allergic rhinitis caused by house dust mite antigen in the U.S. (If house dust mite is positive for MAST ≥ Class 3 or ImmunoCAP® ≥3.5 kUA/L)
  2. Moderate-severe persistent rhinitis when evaluated according to ARIA (Allergic rhinitis and its impact on asthma)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of transcriptomic profiles based on RNA | 4-6 months after baseline
  Based on RNA extracted from skin samples, transcriptomic profiles are analyzed to identify related RNAs that show meaningful changes compared to normal people and immunotherapy using heatmap, and it is estimated that Th2 or Treg-related RNA profiles will be significantly different

SECONDARY OUTCOMES:
Differences in immunological efficacy by type of immunotherapy (subcutaneous, sublingual, percutaneous) | 4-6 months after baseline
  Whether there is a difference in immunological efficacy by type of immunotherapy (subcutaneous, sublingual, percutaneous) is confirmed through pre- and post-group comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hee Park, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided